CLINICAL TRIAL: NCT06357234
Title: A Randomized Controlled Trial Comparing Aprepitant to Standard of Care for Postoperative Nausea and Vomiting Prophylaxis in Children and Adolescents Undergoing Scoliosis Surgery: The APRE-PONV Trial
Brief Title: Aprepitant Treatment to Prevent Postoperative Nausea and Vomiting in Children Undergoing Scoliosis Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: APRE-2023
Record Dates: First submitted 2024-01-17; First posted 2024-04-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-09

CONDITIONS: Spinal Fusion; Nausea and Vomiting, Postoperative; Anesthesia
Keywords: pediatric; anesthetic; scoliosis; Aprepitant
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Scoliosis | interventions — Aprepitant; Glucose

STUDY DESIGN:
Intervention Model Description: This is a randomized double-blind placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment arm of participants will be masked until data collection is complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aprepitant (Experimental): Two doses of 40mg (2ml) Aprepitant
  Interventions: Drug: Aprepitant
- Dextrose (Placebo Comparator): Two doses of dextrose (2ml)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant — Two doses of 40mg (2ml) Aprepitant. One to be given on the morning of surgery and the second on the morning of post-op day 1
  Other Names: Aprepitant oral suspension 20mg/ml
  Arms: Aprepitant
Drug: Placebo — Two doses of dextrose syrup (2ml). One to be given on the morning of surgery and the second on the morning of post-op day 1
  Other Names: Dextrose
  Arms: Dextrose

SUMMARY:
This research trial will measure how useful Aprepitant is in preventing nausea and vomiting in children having surgery to correct scoliosis (curvature of the spine).

DETAILED DESCRIPTION:
Detailed Description: This prospective, randomized, controlled trial will test whether adding Aprepitant to standard multimodal therapy regimen can further reduce the incidence and severity of post-operative nausea and vomiting (PONV) in children undergoing posterior spinal instrumentation and fusion. The primary outcome of the study will be anti-nausea rescue medication administration post-surgery, with secondary outcomes being the first instance of post-surgery anti-nausea rescue medication administration, emesis, headache, flatus, bowel movement, and sensation of itch; incidence of treatment-emergent adverse events; and worst nausea and pain scores post-surgery .

ELIGIBILITY:
Inclusion Criteria:

* Posterior Spinal Instrumentation and Fusion (PSIF) for idiopathic scoliosis
* The fusion must include at least 6 vertebral levels.
* Children greater than or equal to 8 years old, and less than 19 years old on the day of surgery
* Weight > 40kg - for ease of pharmacy preparation (PONV dose 1mg per kg to max 40mg)

Exclusion Criteria:

* Patient/ Parent refusal
* Hypersensitivity to Aprepitant or any ingredient in the formulation or oral solution. (previous allergy or adverse reaction to Aprepitant)
* Developmental delay as reported by parents
* Pregnant - Pregnancy test done as standard of care pre-operative
* Severe systemic disease ASA classification III or greater
* Concurrent use of any medication with severe interaction with Aprepitant as outlined in product monograph.
* Neuromuscular or congenital scoliosis
* Inability to take PO medications

Ages: 8 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Anti-Nausea Rescue Medication | From surgery end-time until discharge, estimated period of up to 10 days
  Anti-nausea rescue medication administered (yes/no).

SECONDARY OUTCOMES:
Anti-nausea rescue medication administered by post-operative day | From surgery end-time until first instance (yes) or until discharge (if no instances during post-operative period),estimated period of up to 10 days
  Anti-nausea rescue medication administered (yes/no). Assessed each post-operative day. The primary outcome is whether nausea rescue medication is used at all in the post-operative period. The secondary outcome is the time (By post operative day) when the first rescue medication is administered.
Emesis (Yes/No) | From surgery end-time until first instance (yes) or until discharge (if no instances during post-operative period), estimated period of up to 10 days
  Assessed each post operative day
Baxter Retching Faces score | From surgery end time until discharge,estimated period of up to 10 days
  Baxter Retching Faces (BARF) scale of nausea - worst score collected twice per post-operative day. Scores range from 0 to 10. Higher scores indicate a worse outcome (0=no nausea at all, 10=the most nausea it is possible to feel).
Pain score | From surgery end time until discharge, estimated period of up to 10 days
  Faces pain scale revised - worst score. Collected twice per post-operative day Faces pain scale-revised: Score of 0 to 10. Higher scores indicate a worse outcome (0=no pain, 10=very much pain).
Headache (yes/no) | From surgery end-time until first instance (yes) or until discharge (if no instances during post-operative period), estimated period of up to 10 days
  Recorded as headache (yes/No) Assessed each post-operative day
Flatus (yes/no) | From surgery end-time until first instance (yes) or until discharge (if no instances during post-operative period), estimated period of up to 10 days
  Assessed each post-operative day
Bowel Motility (yes/no) | From surgery end-time until first instance (yes) or until discharge (if no instances during post-operative period),estimated period of up to 10 days
  Assessed each post-operative day
Sensation of Itch | From surgery end-time until first instance (yes) or until discharge (if no instances during post-operative period),estimated period of up to 10 days
  Assessed each post-operative day
Treatment of emergent adverse events | From administration of first dose of study drug (or placebo) to discharge],estimated period of up to 10 days
  Assessed each day from time of administration of study drug or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Kiberd, MD, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Sciences Center, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Background] Weibel S, Rucker G, Eberhart LH, Pace NL, Hartl HM, Jordan OL, Mayer D, Riemer M, Schaefer MS, Raj D, Backhaus I, Helf A, Schlesinger T, Kienbaum P, Kranke P. Drugs for preventing postoperative nausea and vomiting in adults after general anaesthesia: a network meta-analysis. Cochrane Database Syst Rev. 2020 Oct 19;10(10):CD012859. doi: 10.1002/14651858.CD012859.pub2. PMID 33075160
- [Background] Eberhart LHJ, Geldner G, Kranke P, Morin AM, Schauffelen A, Treiber H, Wulf H. The development and validation of a risk score to predict the probability of postoperative vomiting in pediatric patients. Anesth Analg. 2004 Dec;99(6):1630-1637. doi: 10.1213/01.ANE.0000135639.57715.6C. PMID 15562045
- [Background] Apfel CC, Philip BK, Cakmakkaya OS, Shilling A, Shi YY, Leslie JB, Allard M, Turan A, Windle P, Odom-Forren J, Hooper VD, Radke OC, Ruiz J, Kovac A. Who is at risk for postdischarge nausea and vomiting after ambulatory surgery? Anesthesiology. 2012 Sep;117(3):475-86. doi: 10.1097/ALN.0b013e318267ef31. PMID 22846680
- [Background] Kranke P, Eberhart LH, Toker H, Roewer N, Wulf H, Kiefer P. A prospective evaluation of the POVOC score for the prediction of postoperative vomiting in children. Anesth Analg. 2007 Dec;105(6):1592-7, table of contents. doi: 10.1213/01.ane.0000287816.44124.03. PMID 18042855
- [Background] Aapro M, Carides A, Rapoport BL, Schmoll HJ, Zhang L, Warr D. Aprepitant and fosaprepitant: a 10-year review of efficacy and safety. Oncologist. 2015 Apr;20(4):450-8. doi: 10.1634/theoncologist.2014-0229. Epub 2015 Mar 20. PMID 25795636
- [Background] Salman FT, DiCristina C, Chain A, Afzal AS. Pharmacokinetics and pharmacodynamics of aprepitant for the prevention of postoperative nausea and vomiting in pediatric subjects. J Pediatr Surg. 2019 Jul;54(7):1384-1390. doi: 10.1016/j.jpedsurg.2018.09.006. Epub 2018 Sep 21. PMID 30381138
- [Background] Diemunsch P, Gan TJ, Philip BK, Girao MJ, Eberhart L, Irwin MG, Pueyo J, Chelly JE, Carides AD, Reiss T, Evans JK, Lawson FC; Aprepitant-PONV Protocol 091 International Study Group. Single-dose aprepitant vs ondansetron for the prevention of postoperative nausea and vomiting: a randomized, double-blind phase III trial in patients undergoing open abdominal surgery. Br J Anaesth. 2007 Aug;99(2):202-11. doi: 10.1093/bja/aem133. Epub 2007 May 30. PMID 17540667
- [Background] Gan TJ, Apfel CC, Kovac A, Philip BK, Singla N, Minkowitz H, Habib AS, Knighton J, Carides AD, Zhang H, Horgan KJ, Evans JK, Lawson FC; Aprepitant-PONV Study Group. A randomized, double-blind comparison of the NK1 antagonist, aprepitant, versus ondansetron for the prevention of postoperative nausea and vomiting. Anesth Analg. 2007 May;104(5):1082-9, tables of contents. doi: 10.1213/01.ane.0000263277.35140.a3. PMID 17456656
- [Background] Hasan AME, Abdelzaam E-S. A comparative study between Aprepitant only versus combined ondansetron and Aprepitant as antiemetic therapy, regarding efficacy and duration, in patients undergoing laparoscopic bariatric surgery double-blinded, randomized control clinical trial. J Anesth Clin Res. 2019;10(5)
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Watcha MF, Lee AD, Medellin E, Felberg MT, Bidani SA. Clinical Use of the Pictorial Baxter Retching Faces Scale for the Measurement of Postoperative Nausea in Children. Anesth Analg. 2019 Jun;128(6):1249-1255. doi: 10.1213/ANE.0000000000003850. PMID 31094795